CLINICAL TRIAL: NCT05940272
Title: Evaluation of a Communication Intervention (Hematolo-GIST) for Large B-Cell Lymphoma Providers
Brief Title: Study of a Communication Training Intervention for Large B-Cell Lymphoma Providers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-164
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Lymphoma, B-Cell; Lymphoma; Large-cell Lymphoma; Large B-cell Lymphoma; DLBCL - Diffuse Large B Cell Lymphoma; Mediastinal B-Cell Diffuse Large Cell Lymphoma
Keywords: oncologist; hemotologic oncologist; lymphoma; large cell lymphoma; large b-cell lymphoma; DLBCL; Diffuse Large B Cell Lymphoma; Mediastinal B-Cell Diffuse Large Cell Lymphoma; Hematolo-GIST; 23-164; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hematologists (Experimental): Hematologists will be recruited from the lymphoma clinics at MSK
  Interventions: Behavioral: Hematolo-GIST Training
- Participants Patients (Experimental): Participant patients are being treated by a hematologic oncologist participating in this study
  Interventions: Behavioral: Participants Appointment

INTERVENTIONS:
Behavioral: Hematolo-GIST Training — Hematologist will participate in a group Hematolo-GIST training provided remotely via the study team.
  Arms: Hematologists
Behavioral: Participants Appointment — Participants will meet with Hematolo-GIST trained hematologists. Participants will consent to having their appointment audio-recorded on password-protected devices or MSK approved secure platforms.
  Arms: Participants Patients

SUMMARY:
The purpose of this study is to develop and test a new communication training intervention called Hematolo-GIST to help oncologists communicate with patients about their lymphoma diagnosis and advance care planning.

ELIGIBILITY:
Inclusion Criteria:

Providers

* Currently a an MSK provider caring for patients with DLBCL (including DLBCL-transformed follicular lymphoma (TFL) and primary mediastinal B-cell lymphoma (PMBCL) which are histologically similar and treated as large-cell lymphoma)

Patients

* Per medical record, is currently being treated by a provider who is participating in this study (for the purposes of this study, "treating provider" will be defined as any provider who provides care related to the patient's lymphoma diagnosis)
* Per medical record, has a diagnosis of DLBCL including DLBCL-transformed follicular lymphoma (TFL) and primary mediastinal B-cell lymphoma (PMBCL) which are histologically similar and clinically treated as large-cell lymphoma
* Per medical record, relapse/ refractory disease within 12 months of 4 cycles of first line therapy OR relapse after 2 cycles of later line therapy or or autologous stem cell transplant (ASCT)
* Self-identify as Black and/or White
* Per medical record, 18 years of age or older
* Per self-report, fluent in English**

  * Language verification: Prior to enrollment, patients will be asked the following two questions by a Clinical Research Coordinator (CRC) to verify English fluency necessary for participation in the study:

    1. How well do you speak English? (must respond "very well" or "well" when given the choices of Very well, Well, Not well, Not at all, Don't know, or Refused)
    2. What is your preferred language for healthcare? (must respond English)

Exclusion Criteria:

Providers

* Per self-report, planning to leave the cancer center in the next 12 months

Patients

* Cognitively impaired as demonstrated by (Blessed Orientation- Memory- Concentration (BOMC) score of ≥ 11
* Per research staff judgment and/or self-report, too ill or weak to complete study procedures
* Per medical record or self-report, receiving hospice care at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2028-07-03 (Estimated); Study Completion 2028-07-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Hematolo-GIST intervention among hematologists and participants | Up to 1 year
  Feasbility is defined as ≥70% of screened eligible hematologists and participants enrolling in the study and ≥80% of hematologists learning the approach

CONTACTS AND LOCATIONS:
Overall Officials: Kelly McConnell, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center (All protocol activities), New York, New York
  - NEW YORK PRESBYTERIAN HOSPITAL (Data Collection Only), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org